CLINICAL TRIAL: NCT02484248
Title: Double-blind, Placebo-controlled, Cross-over Trial of Ketotifen in Children and Adolescents With Functional Dyspepsia in Association With Duodenal Eosinophilia
Brief Title: Ketotifen for Children With Functional Dyspepsia in Association With Duodenal Eosinophilia
Acronym: Ketotifen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Craig A. Friesen, MD (Other)
Responsible Party: Sponsor-Investigator, Craig A. Friesen, MD, Division Chief Gastroenterologist, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14110467
Record Dates: First submitted 2015-01-13; First posted 2015-06-29 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Functional Dyspepsia
Keywords: pediatric; eosinophilia; duodenal; ketotifen; functional dyspepsia
MeSH Terms: conditions — Eosinophilia | interventions — Ketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cross-over of Ketotifen (Active Comparator): Patients will begin the active ketotifen treatment first and cross over to placebo.
  Interventions: Drug: Ketotifen
- cross-over of Placebo (Placebo Comparator): Patients will begin the placebo treatment first and cross over to the active ketotifen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketotifen — Ketotifen is an anti-histamine approved by the U.S. FDA to prevent and treat itching of the eyes caused by allergies.
  Arms: cross-over of Ketotifen
Drug: Placebo — The placebo tablet looks identical to the ketotifen tablet, but does not contain ketotifen.
  Arms: cross-over of Placebo

SUMMARY:
Acid reduction remains the most common treatment prescribed empirically by pediatric gastroenterologists for children with functional dyspepsia (FD). When acid reduction therapy fails to provide patients with a therapeutic effect, ketotifen and cromolyn, mast cell stabilizers, represent an attractive potential therapy given data implicating mast cells in the generation of dyspeptic symptoms. Although there have been no adult or pediatric studies on the use of mast cell stabilizers in patients with FD, benefit has been demonstrated in adults with IBS and children with eosinophilic gastroenteritis. Additionally, previous studies show mucosal eosinophilia is highly correlated with functional dyspepsia. Our usual current treatment pathway for functional dyspepsia in association with duodenal mucosal eosinophilia is as follows: acid-reducing medication/montelukast → addition of H1 antagonist → addition of budesonide → addition of oral cromolyn. If ketotifen is effective, it offers the advantage of being able to replace both the H1 antagonist and the oral cromolyn at a substantially reduced cost (approximately 10% of the cost of cromolyn alone). This study aims to introduce ketotifen earlier in the treatment pathway to examine its efficacy on children with functional dyspepsia in association with duodenal eosinophilia.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, cross-over trial of ketotifen in children ages 8 through 17 inclusive that have a diagnosis of functional dyspepsia and have had continued abdominal pain despite acid reduction therapy in combination with montelukast. The primary aim is to assess the symptomatic response to ketotifen as compared to placebo in children with functional dyspepsia in association with duodenal eosinophilia who have previously had worsening, no clinical change, or only a partial response to acid-reduction therapy in combination with montelukast.

The study lasts 147 days for subjects responsive to ketotifen and 63 days for those who are not. For those who respond to ketotifen, there are 4 clinic visits and 3 phone interviews. Clinic visits include a physical, blood draws, questionnaires, review of medical history and medications; phone interviews involve answering a few questions. For those who do not respond to ketotifen, there are 3 clinic and 2 phone visits. Subjects who enroll in the study are randomly assigned to Group A or Group B. The subject, subject's parents, and study staff will not know to which group the subject is assigned. Group A will be given a placebo, an inactive pill with no medication in it, for days 1-28, and switched to ketotifen for days 36-63. Group B will be given ketotifen for days 1-28 and switched to placebo for days 36-63. The group assignment will be unblinded at day 63, at which point initial ketotifen responders will undergo an open-label twelve week trial of ketotifen to assess sustainability.

Secondary aims include: 1) assessing the impact of ketotifen as compared to placebo on quality of life; 2) assessing the sustainability of response to ketotifen in initial responders, and 3) assessing the pharmacokinetics of ketotifen in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 8 and 17 years, inclusive
2. abdominal pain of at least 8 weeks duration and fulfilling symptom-based criteria for functional dyspepsia(5);
3. previous endoscopy with biopsies demonstrating >20 eosinophils/high powered field on duodenal mucosal biopsies;
4. previous treatment with acid-reduction therapy and montelukast with a level 3 (as defined below)or lesser response;
5. evidence of written parental permission (consent) and subject assent;
6. Negative pregnancy screening for females of child bearing potential.

Exclusion Criteria:

1. previous treatment with ketotifen;
2. treatment with oral corticosteroids or oral cromolyn sodium in the 6 months prior to enrollment;
3. any prior history of diabetes mellitus, cancer, chronic cardiac disease, respiratory disease, or renal disease requiring routine medical care;
4. Pregnant/planning to become pregnant;
5. Post-menarche females unwilling to use highly-efficacious contraception to prevent pregnancy;
6. Epilepsy or history of seizures;
7. Liver disease or elevation of liver enzymes;
8. Use of oral hypoglycemic medications, antipsychotics, benzodiazepines, tricyclic antidepressants, barbiturates, or opioids;
9. Allergy to ketotifen or other products in capsule
10. Refusal of Urine pregnancy test in post-menarchal females.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete Physical | day 0, day 28, day 63, and day 147
  The study physician will check all systems and ask questions about pain and symptoms. This is a comprehensive system check to ensure safety. Change is assessed from each time period.
Blood pressure | day 0, day 28, day 63, and day 147
  A trained professional will measure blood pressure to ensure value is within normal range and ensure safety of patient. Change is assessed from each time period.
Liver Functioning Test (a test ran from a blood sample to check a patients liver functioning) | day 0, day 28, day 63, and day 147
  A blood sample is collected and tested by a certified laboratory for liver function. This will be completed and verified to be within normal ranges by the study physician to ensure patient safety. Change is assessed from each time period.
State-Trait Inventory for Cognitive and Somatic Anxiety - Child Version | day 0, day 28, day 63, and day 147
  Anxiety score testing assessed with questionnaires. Anxiety scores are correlated with pain. Change is assessed from each time period.
Pediatric Quality of Life Inventory | day 0, day 28, day 63, and day 147
  Quality of life survey for pediatrics to ensures maintenance of quality of life throughout study. Change is assessed from each time period.
Heart Rate | day 0, day 28, day 63, and day 147
  A trained professional will measure heart rate to ensure value is within normal range and patient safety. Change is assessed from each time period.
Respiratory Rate | day 0, day 28, day 63, and day 147
  A trained professional will measure respiratory rate to ensure value is within normal range and patient safety. Change is assessed from each time period.

SECONDARY OUTCOMES:
Pharmacokinetic Sampling (Area under the plasma concentration versus time curve - AUC) | day 0, day 28, day 63, and day 147
  Pharmacokinetic sampling allows for evaluation of the entire process of the drug breakdown by the body and ensures long term efficacy and safety. Change is being assessed from each time period.
Pharmacokinetics Sampling (Peak Plasma Concentration - Cmax) | day 0, day 28, day 63, and day 147
  Pharmacokinetic sampling allows for evaluation of the entire process of the drug breakdown by the body and ensures long term efficacy and safety. Change is being assessed from each time period.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Friesen, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] McFadyen ML, Miller R, Ludden TM. Ketotifen pharmacokinetics in children with atopic perennial asthma. Eur J Clin Pharmacol. 1997;52(5):383-6. doi: 10.1007/s002280050305. PMID 9272408
- [Background] Klooker TK, Braak B, Koopman KE, Welting O, Wouters MM, van der Heide S, Schemann M, Bischoff SC, van den Wijngaard RM, Boeckxstaens GE. The mast cell stabiliser ketotifen decreases visceral hypersensitivity and improves intestinal symptoms in patients with irritable bowel syndrome. Gut. 2010 Sep;59(9):1213-21. doi: 10.1136/gut.2010.213108. Epub 2010 Jul 21. PMID 20650926
- [Background] Schurman JV, Singh M, Singh V, Neilan N, Friesen CA. Symptoms and subtypes in pediatric functional dyspepsia: relation to mucosal inflammation and psychological functioning. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):298-303. doi: 10.1097/MPG.0b013e3181d1363c. PMID 20479684
- [Background] Hall W, Buckley M, Crotty P, O'Morain CA. Gastric mucosal mast cells are increased in Helicobacter pylori-negative functional dyspepsia. Clin Gastroenterol Hepatol. 2003 Sep;1(5):363-9. doi: 10.1053/s1542-3565(03)00184-8. PMID 15017654
- [Background] Friesen CA, Lin Z, Singh M, Singh V, Schurman JV, Burchell N, Cocjin JT, McCallum RW. Antral inflammatory cells, gastric emptying, and electrogastrography in pediatric functional dyspepsia. Dig Dis Sci. 2008 Oct;53(10):2634-40. doi: 10.1007/s10620-008-0207-0. Epub 2008 Mar 5. PMID 18320315
- [Background] Friesen CA, Neilan NA, Schurman JV, Taylor DL, Kearns GL, Abdel-Rahman SM. Montelukast in the treatment of duodenal eosinophilia in children with dyspepsia: effect on eosinophil density and activation in relation to pharmacokinetics. BMC Gastroenterol. 2009 May 11;9:32. doi: 10.1186/1471-230X-9-32. PMID 19432972
- [Background] Santos J, Saperas E, Nogueiras C, Mourelle M, Antolin M, Cadahia A, Malagelada JR. Release of mast cell mediators into the jejunum by cold pain stress in humans. Gastroenterology. 1998 Apr;114(4):640-8. doi: 10.1016/s0016-5085(98)70577-3. PMID 9516384
- [Background] Stefanini GF, Saggioro A, Alvisi V, Angelini G, Capurso L, di Lorenzo G, Dobrilla G, Dodero M, Galimberti M, Gasbarrini G, et al. Oral cromolyn sodium in comparison with elimination diet in the irritable bowel syndrome, diarrheic type. Multicenter study of 428 patients. Scand J Gastroenterol. 1995 Jun;30(6):535-41. doi: 10.3109/00365529509089786. PMID 7569760
- [Background] Chen X, Zhong D, Liu D, Wang Y, Han Y, Gu J. Determination of ketotifen and its conjugated metabolite in human plasma by liquid chromatography/tandem mass spectrometry: application to a pharmacokinetic study. Rapid Commun Mass Spectrom. 2003;17(22):2459-63. doi: 10.1002/rcm.1189. PMID 14608613
- [Background] Grahnen A, Lonnebo A, Beck O, Eckernas SA, Dahlstrom B, Lindstrom B. Pharmacokinetics of ketotifen after oral administration to healthy male subjects. Biopharm Drug Dispos. 1992 May;13(4):255-62. doi: 10.1002/bdd.2510130404. PMID 1600111
- [Derived] Friesen CS, Shakhnovich V, Toren P, Retke B, Schurman J, Colombo J, Deacy A, Friesen CA, Abdel-Rahman S. A Pilot Study of Ketotifen in Patients Aged 8-17 Years with Functional Dyspepsia Associated with Mucosal Eosinophilia. Paediatr Drugs. 2024 Jul;26(4):451-457. doi: 10.1007/s40272-024-00628-8. Epub 2024 May 21. PMID 38771467